CLINICAL TRIAL: NCT07344805
Title: Clinical Effects and Metagenomic Analysis of Using an Air Polishing Device With Erythritol Powder Compared to Scaling and Root Planing in Periodontal Maintenance Therapy: A Randomized Clinical Trial
Brief Title: Clinical Effects and Metagenomic Analysis of Using an Air Polishing Device With Erythritol Powder Compared to Scaling and Root Planing in Periodontal Maintenance Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Chirag Sheth, Associate Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEU-Martinez-Gonzalez-Cortell
Record Dates: First submitted 2025-11-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis
Keywords: periodontal maintenance; erythritol; powder air polishing
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontal maintenance with ultrasonic + scaling and root planning (Active Comparator)
  Interventions: Device: Cavitron® ultrasonic scaler
- Periodontal maintenance with erythritol air polishing (Experimental)
  Interventions: Device: AIRFLOW® Prophylaxis Master

INTERVENTIONS:
Device: AIRFLOW® Prophylaxis Master — Periodontal Maintenance with Erythritol Air Polisher in periodontal patients.
  Arms: Periodontal maintenance with erythritol air polishing
Device: Cavitron® ultrasonic scaler — Periodontal maintenance with ultrasonic scaler and manual curettes in periodontal patients.
  Arms: Periodontal maintenance with ultrasonic + scaling and root planning

SUMMARY:
Periodontitis is a chronic, multifactorial disease primarily driven by the accumulation of bacterial deposits. Treatment involves the mechanical removal of the biofilm, traditionally performed by scaling and root planing (SRP). However, SRP is time-consuming and can cause irreversible damage to both hard and soft tissues as well as postoperative sensitivity. Consequently, adjunctive or alternative air-polishing devices have been developed. The objective of this study is to compare the clinical and microbiological efficacy of an erythritol-powder air-polishing device versus SRP in periodontal maintenance therapy.To evaluate patient-reported pain and treatment time for erythritol air-polishing versus SRP. A randomized clinical trial was designed and participants were randomly assigned to one of two groups: Intervention: Perio-Flow® (air + erythritol powder) and PIEZON PS®. Control: Ultrasonic debridement followed by SRP with Gracey curettes.At baseline and at six months, probing depth, clinical attachment level, and bleeding on probing were recorded. Saliva samples were collected to detect the most prevalent periodontal pathogens. Patient discomfort during treatment was measured by a visual analog scale, and procedure duration was timed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received basic periodontal treatment between 3-6 months before the study.

Exclusion Criteria:

* Pregnant or breastfeeding patients.
* Use of systemic antibiotics within 6 months prior to the study.
* Patients who smoke more than 10 cigarettes/day.
* Uncontrolled diabetic patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Improvement of clinical periodontal parameter: clinical attachment level | six months
  Measurement of clinical attachment level in milimeters
Improvement of clinical periodontal parameter: probing depth | six months
  Measurement of probing depth in milimeters
Improvement of clinical periodontal parameter: bleeding index | six months
  Measurement of bleeding index in percentage.

SECONDARY OUTCOMES:
Changes in periodontal microbiome | Six months
  We will present the following analyses:
  * Overall and differential abundance
  * Comparative relative inter-group community structure differences
  The overall and differential abundance of taxa will be analyzed using Kruskal Wallis non-parametric test. FDR Benjamini-Hochberg correction will be used to correct for multiple comparisons.
  Differences in community structure between experimental and control groups will be tested using Permanova. Permdisp test will be used to identify location vs. dispersion effects .
  The threshold for significance for all analyses will be set at p ≤ 0.05.
  'BiodiversityR' version 2.11-1, 'PMCMR' version 4.3 and 'vegan' version 2.5-5 packages of the R software package version 36.6.0 (www.R-project.org) will be used.

OTHER OUTCOMES:
Patient discomfort | Six months
  Measurement of patient discomfort during the treatment by Visual Analogue Scale (VAS) Questionnaire (from no pain (score 0) to maximum pain imaginable (score 7)).

CONTACTS AND LOCATIONS:
Overall Officials: Isidoro Cortell-Ballester, DDS, MD, PhD, Study Director — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No